CLINICAL TRIAL: NCT06490770
Title: Analysis of the Pathophysiological and Functional State of the Knee Joint
Acronym: Gait-MRI-Knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Gait-MRI-Knee
Record Dates: First submitted 2024-06-13; First posted 2024-07-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Knee; Cartilage Degeneration
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Gait Analysis; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- group 1 (Other)
  Interventions: Diagnostic Test: Gait analysis, Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Gait analysis, Magnetic Resonance Imaging — Gait analysis and Magnetic Resonance Imaging to investigate the functionality and the pathological condition of the knee, respectively

SUMMARY:
Osteoarthritis is the most common degenerative condition affecting the knee joint globally, with an incidence of about 7% of the population. In Italy, it affects approximately 3.9 million people, with a direct treatment cost of around €2.5 billion. At the joint level, osteoarthritis manifests with pain and reduced functionality, worsening as the disease progresses and severely limiting knee movement. Compounding this, osteoarthritis can impact both elderly and younger individuals due to traumatic factors.

Despite its significant impact, effective treatments for osteoarthritis that address its underlying causes are still lacking, focusing mainly on symptom management. Therefore, improving diagnostic and prognostic approaches is crucial to better understand its onset and progression.

MRI is a primary diagnostic tool for assessing the knee joint's pathophysiological state. It uses tissue-specific sequences to investigate joint homeostasis in detail, although it primarily provides insights into morphology, structure, and tissue composition rather than functional changes within the joint. This limitation is noteworthy because joint homeostasis involves complex interactions among biomechanical, structural, and biological processes, which are directly influenced by osteoarthritis.

Gait analysis provides valuable diagnostic information on joint function. By integrating sensor measurements and electronic systems with patient-specific musculoskeletal models derived from MRI morphometric data, it is possible to assess the forces and moments within the joint during specific movements.

Given that osteoarthritis affects the entire joint, employing multidisciplinary approaches can enhance diagnostic precision and provide insights into the progressive impact of degenerative conditions like osteoarthritis on joint health.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain and/or loss of functionality
* Kellgren-Lawrence grade less than or equal to 2
* Arthroscopic evidence of cartilage tissue lesions
* Evidence of cartilage and/or meniscal tissue degeneration and/or subchondral bone marrow lesions

Exclusion Criteria:

* History/evidence of previous partial or total knee prosthesis interventions
* Inability to provide informed consent
* Conditions or physical disorders incompatible with the use of MRI and electrical stimulation (implanted active and passive biomedical devices, epilepsy, severe venous insufficiency in the lower limbs)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging | at baseline and 12-month follow-up
  MRI images will be acquired for each subject using a high-field scanner (3T, Discovery MR750w3, GE Healthcare, UK) with sequences that will allow i) the analysis of the pathophysiological state of the knee cartilage, and ii) the identification and segmentation of the various leg muscles.
  Regarding the investigation of joint tissues, quantitative sequences (e.g., T2 mapping) will be acquired using a specific coil, according to standard practice. MRI images related to the muscular aspects of the entire lower limb will be added to the previous ones-which will instead be focused on the region bounded by the femoral and tibial diaphyses-in order to obtain complete information in a single acquisition session with additional timing on the order of minutes. MRI images at the 12-month follow-up are specific to the study.

SECONDARY OUTCOMES:
Strength measurements with a manual dynamometer | at baseline and 12-month follow-up
  As per clinical practice, before gait analysis, muscle strength (generalized, not specific to the knee flexor and extensor muscles) will be measured through the execution of a hand grip test with a manual hydraulic dynamometer (Jamar, Sammons Preston Rolyan, USA). The measurement will be repeated three times, allowing a 1-minute rest between repetitions.
Bioimpedance analysis | at baseline and 12-month follow-up
  Patients will be asked to undergo a bioimpedance measurement (BIA BIVA 101 PRO, Akern, ITA) to estimate the muscle mass (residual) and fat mass for both lower limbs.
Gait Analysis (including Electromyography) | at baseline and 12-month follow-up
  Gait analysis with electromyographic signal acquisition will be performed. Anthropometric measurements will be taken, and retroreflective markers will be placed on anatomical landmarks. Bipolar electrodes will be positioned on key lower limb muscles according to SENIAM guidelines. The test includes static calibration, walking, sit-to-stand-to-sit, and step-over tasks. Electromyographic signals will be monitored and analyzed for muscle activation and co-activation. The session will last 40-60 minutes and is study-specific.
Clinical questionnaires | at baseline and 12-month follow-up
  Knee function and pain will be assessed using the WOMAC (Western Ontario and McMaster Universities Arthritis Index) and KOOS (Knee Injury and Osteoarthritis Outcome Score) scales. WOMAC is a self-assessment questionnaire with 24 questions divided into three subgroups evaluating knee pain, joint stiffness, and functionality during daily activities. KOOS evaluates symptoms, pain, daily activities, sports activities, and quality of life.
  A dedicated data collection form will be used to gather all clinical information and study results. For each patient, a paper Case Report Form (CRF) will be completed. Additionally, all collected experimental data will be saved in a specially created folder on the Institute's secure server.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy